CLINICAL TRIAL: NCT05254899
Title: Anti-PD-1 Antibody and P-GEMOX Chemotherapy Combined With Radiotherapy in High-risk Early-Stage Extranodal NK/T Cell Lymphoma, Nasal Type: A Multi-center Phase II Study
Brief Title: Anti-PD-1 Antibody and P-GEMOX Chemotherapy Combined With Radiotherapy in High-risk Early-Stage ENKTL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); The Affiliated Hospital Of Guizhou Medical University (Other); The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Shunan Qi, Associated Prof. in the radiation oncology department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCG-NKT-2102
Record Dates: First submitted 2021-11-07; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Extranodal NK-T-Cell Lymphoma, Nasal and Nasal-Type; Early-stage; High-Risk Cancer
Keywords: NK/T-Cell Lymphoma, Nasal and Nasal-Type; anti-PD-1 antibody; radiotherapy; chemotherapy; Pegaspargase
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — spartalizumab; tislelizumab; pegaspargase; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inductive and concurrent anti-PD-1 antibody combined with chemo-radiotherapy (Experimental): All the enrolled patients receive 3 cycles of anti-PD-1 antibody (Tislelizumab 200mg d1) + P-GEMOX (Pegaspargase 3000u d2, Gemcitabine 1g/m2 d2, Oxaliplatin 85mg/m2 d2) systemic treatment every 14 days, followed by involved-site radiotherapy with concurrent anti-PD-1 antibody (Tislelizumab 200mg) every two weeks.
  Interventions: Drug: Anti-PD-1 monoclonal antibody; Drug: Pegaspargase; Drug: Gemcitabine; Drug: Oxaliplatin; Radiation: Involved site radiotherapy

INTERVENTIONS:
Drug: Anti-PD-1 monoclonal antibody — 200mg iv on Day 1 of each 14-day cycle for 3 cycles in induction treatment; 200mg iv on Day 1,15, 29 during RT treatment
  Other Names: Tislelizumab
Drug: Pegaspargase — 3000 U/m2 im on Day 2 of each 14-day cycle for 3 cycles in induction treatment
Drug: Gemcitabine — 1g/m2 iv on Day 2 of each 14-day cycle for 3 cycles in induction treatment
Drug: Oxaliplatin — 1g/m2 iv on Day 2 of each 14-day cycle for 3 cycles in induction treatment
Radiation: Involved site radiotherapy — Involved site radiotherapy according to the ILROG guideline with primary tumor dose of 50-56Gy 14-28 days after inductive therapy

SUMMARY:
The current study is a phase II multi-center single arm trial to evaluate the efficacy and safety of inductive Anti-PD-1+P-GEMOX treatment followed by radiotherapy and concurrent Anti-PD-1 antibody in early-stage high-risk extranodal NK/T cell lymphoma, nasal type

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proved extranodal NK/T cell lymphoma
* No previous anti-cancer treatment
* Measurable lesion on baseline PET/CT and MRI
* Stage I-II
* Have at lest one following risk factor: Elevated serum LDH level; PTI+; stage II
* ECOG PS 0-1
* Sufficient organ functions

Exclusion Criteria:

* Other mature T- or NK- lymphoma
* Hemophagocytic lymphohistiocytosis
* Primary CNS lymphoma or CNS-involved lymphoma
* History of malignancy except for cutaneous basal-/squamous- cell carcinoma or cervical carcinoma in situ 3 years prior to study treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete Response rate after 3 cycles of Anti-PD-1 antibody and P-GEMOX therapy | At the end of Cycle 3 (each cycle is 14 days)
  To evaluate the complete response (CR) rate after 3 cycles of Anti-PD-1 antibody and P-GEMOX therapy according to Lyric 2016 criteria

SECONDARY OUTCOMES:
Progression-free survival rate at year 2 after enrollment, 2y-PFS | 2 year
  From enrollment to disease progression or any death
Overall Survival rate at year 2/5 after enrollment，2y-/5y-OS | 2-year, 5-year
  From enrollment to death
acute toxicity | From enrollment to 3 months after treatment
  evaluated according to the CTCAE criteria
Quality of Life，QoL | baseline, 1/3/6/12/24 months after treatment
  evaluated according to EORTC-QLQ-HN35
Quality of Life，QoL | baseline, 1/3/6/12/24 months after treatment
  evaluated according to EORTC-QLQ-C30

OTHER OUTCOMES:
biomarkers (single cell transcriptomics) | baseline, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shunan M Qi, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided